CLINICAL TRIAL: NCT02188394
Title: Effects of Anesthetic Blockades on Pain Modulation in Migraine
Brief Title: Anesthetic Blockades and Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: César Fernández-de-las-Peñas (Other)
Responsible Party: Sponsor-Investigator, César Fernández-de-las-Peñas, Proffesor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCSC11/263
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Migraine; Pain
Keywords: migraine,; pressure pain,; anesthetic blocks; patients
MeSH Terms: conditions — Pain; Migraine Disorders | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anesthetic blockades with bupivacaine (Experimental): Patients will receive a bilateral greater occipital nerve blockade with bupivacaine 0,5%
  Interventions: Drug: Anesthetic blockades with bupivacaine
- Isotonic saline injection (Placebo Comparator): Patients will receive a bilateral occipital injection with isotonic saline
  Interventions: Drug: Isotonic saline injection

INTERVENTIONS:
Drug: Anesthetic blockades with bupivacaine
  Arms: Anesthetic blockades with bupivacaine
Drug: Isotonic saline injection
  Arms: Isotonic saline injection

SUMMARY:
Greater occipital nerve (GON) anesthetic blockades are widely used for the treatment of headaches, yet its efficacy in migraine has hardly been assessed with controlled studies. The aim of this study is to evaluate the short-term clinical efficacy of GON anaesthetic blockades in chronic migraine and to analyze their effect on pressure pain thresholds (PPTs) in different areas. We hypothesize that those patients receiving real GON anesthetic blockade will receive greater improvements in pain nociception. We will conduct a double-blind, randomized, parallel and placebo-controlled clinical trial where one group will be treated with bilateral GON blockade with bupivacaine 0,5% and the other group will be treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine

Exclusion Criteria:

* Other primary headaches
* Other secondary headaches
* Co-morbid medical diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in the number of days with moderate/intense migraine | Baseline (1 week before) and 1 week after intervention
  A headache diary will register the number of days with moderate/intense migraine. Moderate/intense migraine is considered a headache with an intensity level over 4 points on a numerical pain rate scale (NPRS, 0-10)

SECONDARY OUTCOMES:
Changes in the number of days with mild/moderate migraine | Baseline (1 week before) and 1 week after intervention
  A headache diary will register the number of days with mild/moderate migraine. Moderate/intense migraine is considered a headache with an intensity level under 4 points on a numerical pain rate scale (NPRS, 0-10)
Changes in the number of symptomatic medication drugs | Baseline (1 week before) and 1 week after intervention
  The subjects will register in the headache diary the number of days per week in which they need symptomatic medical drugs for relief the headache attack
Changes in pressure pain thresholds | Baseline, 1 hour after and 1 week after intervention
  Pressure pain thresholds will be assessed over the supraorbital, infraorbital and mental nerves, and over the second metacarpal and tibialis anterior muscle

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luz Cuadrado, MD; PhD, Principal Investigator — Hospital Clinico San Carlos-Universidad Complutense de Madrid
Locations (1):
- Hospital Universitario Clinico San Carlos-Universidad Complutense de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Cuadrado ML, Aledo-Serrano A, Navarro P, Lopez-Ruiz P, Fernandez-de-Las-Penas C, Gonzalez-Suarez I, Orviz A, Fernandez-Perez C. Short-term effects of greater occipital nerve blocks in chronic migraine: A double-blind, randomised, placebo-controlled clinical trial. Cephalalgia. 2017 Aug;37(9):864-872. doi: 10.1177/0333102416655159. Epub 2016 Jun 12. PMID 27296456